CLINICAL TRIAL: NCT03066817
Title: A Pilot Study of Role of Vitamin D in Regulation of Bone Homeostasis in Orthopaedic Polytrauma Patients
Brief Title: Vitamin D and Bone Homeostasis in Ortho Polytrauma Patients
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Waiting for annual IRB progress report to be reviewed and approved
Sponsor: New York City Health and Hospitals Corporation (Other)
Collaborators: Foundation of Orthopedic Trauma (Other); Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSMB01
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Vitamin D Deficiency; Polytrauma; Orthopedic Disorder
Keywords: Vitamin D; Deficiency; Insufficiency; Bone turnover; Bone healing; Polytrauma
MeSH Terms: conditions — Vitamin D Deficiency; Multiple Trauma; Musculoskeletal Diseases | interventions — Ergocalciferols; Fluid Therapy; Propylene Glycol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vitamin D control (Placebo Comparator): The control cohort will receive 50cc of propylene glycol as placebo via oral, nasogastric tube, or gastrostomy route on hospital admission.
  Interventions: Drug: Propylene Glycol
- Vitamin D intervention cohort (Experimental): The intervention cohort will receive a one-time 400,000 IU liquid ergocalciferol (50cc of Ergocalciferol 8000 IU/ML Oral Liquid [DRISDOL]) via oral, nasogastric tube, or gastrostomy route on hospital admission.
  Interventions: Drug: Ergocalciferol 8000 IU/ML Oral Liquid [DRISDOL]

INTERVENTIONS:
Drug: Ergocalciferol 8000 IU/ML Oral Liquid [DRISDOL] — 50cc of ergocalciferol 8000 IU/ml will be given to participants as a one-time dose.
  Other Names: Calcidol
  Arms: Vitamin D intervention cohort
Drug: Propylene Glycol — 50cc of propylene glycole will be given to participants as one-time dose, used as placebo
  Arms: Vitamin D control

SUMMARY:
Although vitamin D is known to play a major role in multiple organ functions in healthy adults, including bone homeostasis, its role in the unique population of orthopaedic polytrauma patients has not been well described. The aim of this therapeutic randomized placebo-controlled feasibility study is to determine the effect of vitamin D supplementation initiated on admission on patients' 25(OH)-D level, bone turnover markers, and clinical outcomes in a cohort of adult orthopaedic polytrauma patients. Polytrauma patients with one or more orthopaedic injuries admitted to an urban Level I trauma center will be screened for eligibility based upon strict inclusion and exclusion criteria. Sixty patients meeting the criteria will be consented, enrolled and randomized in a 1:1 ratio to intervention and control (placebo) arm. Baseline 25(OH)-D and bone turnover marker levels will be drawn for all the patients on admission, and the intervention arm will receive a one-time dose of ergocalciferol (Vitamin D2) 400,000 IU shortly after enrollment. The labs will be repeated 7 days after the initial draw or at discharge, whichever occurs first. Patients' daily immobilization status, baseline characteristics and clinical outcomes will be recorded. Statistical methods will be used to assess whether there is a difference in 25(OH)-D and bone turnover markers levels associated with the intervention.

DETAILED DESCRIPTION:
Sixty polytrauma patients presenting to Jacobi Medical Center will be screened for eligibility according to strict inclusion and exclusion criteria by study personnel on admission. Medical history, physical examination, and laboratory findings will be collected and assessed to ensure that patients meet the inclusion and exclusion criteria. Eligible subjects will be enrolled after obtaining informed consent from either the subject or health care proxy if the subject is not able to participate in the decision-making process secondary to his injuries or mental status. As this dose of vitamin D has not been previously studied in pregnant subjects, female subjects will be counseled on potential pregnancy risks and will undergo urine pregnancy testing prior to administration of the investigational agent/placebo. Female patients testing positive for pregnancy will be removed from the study. Upon enrollment, study personnel will assign subjects a study ID and record this information in a password-protected data collection document.

All enrolled subjects will have blood draws by phlebotomy or nursing staff for the above-mentioned bone turnover markers once consent is obtained. This will include specimen collection and processing for the following serum levels in both study arms: 25(OH)-D, PTH, collagen type I C-telopeptide, calcium, phosphorus, osteocalcin, and alkaline phosphatase. This initial specimen collection will occur in the interval between 0 and 72 hours of hospital admission.

Collected specimen will be assigned unique identifiers corresponding to patients' study IDs and delivered to core labs at Jacobi Medical Center. From there, the specimen will be sent to an outside testing facility (Northwell Laboratories, Lake Success, NY), where specimen processing will occur. Normal laboratory values will be established by the outside testing facility according to CLIA standards.

The study personnel will liaise with the JMC Main or Satellite Pharmacy to alert them regarding newly enrolled study subjects. The pharmacist will then assign patients according to randomization algorithm in a 1:1 ratio to intervention and control arms, with 30 patients in each group by the end of the study accrual. The pharmacist will then prepare and transport the investigational agent or placebo to the subject's location for administration by nursing staff.

The intervention cohort will receive 400,000IU liquid ergocalciferol (50cc of 8000IU/cc Calcidol solution) via oral, NG tube, or gastrostomy route.

The control cohort will receive 50cc of propylene glycol as placebo via oral, NG tube, or gastrostomy route.

A repeat specimen collection of above-mentioned bone turnover markers will commence either at 7 days if patient is still inpatient, or at discharge, whichever occurs first. The specimens obtained at that time will be treated in the same manner as the initial specimens.

For each enrolled subject, the investigators will collect data from hospital presentation to discharge on standard demographics, routine laboratory results, clinical and injury characteristics and hospital course data (length of stay, in-hospital mortality, mobilization status, associated inpatient procedures and complications).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age 18-65 years
2. One or more orthopaedic injuries on admission
3. Admission injury severity score (ISS)≥16
4. Anticipated stay in hospital of more than 7 days

Exclusion Criteria:

1. Pregnancy (if patient becomes pregnant during the study, she will be removed from the study)
2. End stage kidney disease
3. Patients on furosemide, thiazide, or corticosteroid therapy
4. Patients with chronic liver disease
5. Patients with recent history of vitamin D supplementation more than 5000 IU/day
6. Patients actively undergoing chemo- or immunotherapy
7. Patients with hematologic and solid malignancies
8. Patients receiving treatment for osteoporosis
9. Patients with "nothing per mouth" status secondary to any preceding procedures involving their GI system (e.g. patients with colectomy performed on this admission secondary to gunshot wound to abdomen)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
25(OH)-D serum level in relation to other serum markers of bone turnover | 1 week
  Serum Vitamin D Level, Serum Parathyroid Hormone Level, Serum C-terminal Telopeptide Level, Serum Osteocalcin Level

SECONDARY OUTCOMES:
Hospital length of stay | 1 week
  Patient hospital length of stay if patient leaves before hospital day 7
In-hospital morbidity and mortality | 1 week
  Statistics regarding in-hospital morbidity and mortality

CONTACTS AND LOCATIONS:
Overall Officials: Milan Sen, MD, Principal Investigator — Montefiore Medical Center / Jacobi Medical Center
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not planned to be shared.